CLINICAL TRIAL: NCT05727228
Title: Improving Screening Triage in Older Postmenopausal HPV-screen-positive Women Aged 50-64 and Risk-stratification of Women Aged 23-64 After Excision
Brief Title: Screening Triage and Risk Stratification
Acronym: I-share
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Randers Regional Hospital (Other)
Responsible Party: Principal Investigator, Mette Tranberg Nielsen, post doc, PhD, University of Aarhus
Other Study IDs: 2704
Record Dates: First submitted 2023-01-16; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Cervix Cancer; HPV Testing; Postmenopausal Women
Keywords: mass screening; triage biomarkers
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cytological Techniques; DNA Methylation; Viral Load

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cytology, p16/ki67 dual stain cytology (DS), extended genotyping, DNA methylation, viral load, — p16/Ki67 dual stain cytology, extended genotyping and DNA methylation will be performed from the residual cell-pellet from the HPV-positive screening samples. If no cytology-triage testing is performed as a part of the screening algorithm, a cytology will be performed at inclusion. If any residual material is left after DS, extended genotyping and DNA methylation, it will be stores at -80 degrees for future purposes.

SUMMARY:
* To investigate the performance of cytology, extended genotyping, p16/Ki67 dual stain cytology, DNA methylation and viral load as triage markers in post-menopausal HPV-screen-positive women aged 50-64 years in the organized screening program to predict the risk of developing CIN2+. (work package 1)
* To investigate the performance of cytology, extended genotyping, p16/Ki67 dual stain cytology, DNA methylation and viral load six months after cervical excision to predict the long-term risk of residual/recurrent CIN2+ lesions among women aged 23-64 (work-package 2)

DETAILED DESCRIPTION:
As HPV-positive women may have a transient infection which would be cleared with treatment, triage of HPV-positive women are needed to decrease the colposcopy referral. Liquid-based cytology (hereinafter cytology) are often used as triage for HPV-positive women. HPV 16/18 are the predominant HPV types in younger women and are for all aged referred directly for colposcopy. However as women age, hrHPV other types become more prevalent(10) and these types are triaged with cytology. However, as cytology undergo subjective interpretation and as it may have a decreased sensitivity in with increasing age(11, 12) cytology may not be the most optimal triage marker in postmenopausal women.

p16/Ki67 dual stain cytology (hereinafter DS) is another triage marker. p16 is a cell-cycle regulator protein and Ki67 is a proliferation-associated protein which under normal circumstances are mutual exclusive. Thus, in an HPV-transformed cell co-expression of p16 and Ki67 indicates cell deregulation and increased risk of cervical precancer.(13) In several studies DS have shown better sensitivity and negative predictive value (NPV) as compared to cytology in triaging HPV-positive women(14-17) and women with low-grade cytology (ASC-US and LSIL)(18-20).

Methylation of HPV-positive women benefits from a more objective evaluation than both cytology and DS and has in shown promising results in triaging HPV-positive women.(21) Most studies on DS and methylation have however, been conducted in younger women and studies evaluation the performance in postmenopausal women are needed.

Women diagnosed with CIN2+ undergo excisional treatment removing the lesions and thereby reducing the woman's risk of developing cervical cancer. The most frequently used method is loop electrosurgical excision procedure (LEEP). Despite treatment, women previously diagnosed with CIN3+ lesion are at greater risk of developing cervical cancer with the risk increasing with increasing age.(22) Surveillance after LEEP consist of test-of cure (i.e. cytology and HPV test) six months after LEEP in several countries.(23-27) Treatment of CIN2+ is however, not always successful and residual or recurrent high-grade disease (CIN2+) occurs on average in 8% (ranging from 4% to 18%) of treated women, with the majority of treatment failure occurring mainly the first two post-operative years.(28, 29) Persistent HPV infection and positive margins after LEEP are risk factors for residual or recurrent disease after LEEP(28). However, not all women are at the same risk of recurrent disease, but still managed the same way as women at higher risk and therefore a future risk-stratification are needed to individualize the follow-up pathways. Moreover, introduction of a risk-stratification in the follow-up pathway may also decrease the number of open-ended follow-up pathways. In a recent study in HPV-positive women 60-64 years only 26% had follow-up as recommended.(30)

ELIGIBILITY:
Inclusion Criteria:

* HPV-screen-positive (aged 50-64)
* Women who undergo test-of-cure (i.e. HPV and cytology) six months after LEEP in Central Denmark Region (aged 23-64)
* Women who undergo follow-up test (i.e. HPV and cytology) 12 months after LEEP
* A valid cytology-triage result (aged 23-64)

Exclusion Criteria:

* Listed in the registry as a person who have rejected to participate in research
* Invalid cytology and HPV result six months after LEEP
* No residual material available

Ages: 23 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is focused on cervical cancer screening and as only women had a cervix, only women will be included in this study.
Study Population: Women aged 50-65 who have been tested HPV-screen positive
  Women aged 23-64 who undergo test-of-cure or follow-up test after LEEP
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-02-27 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The number of women with CIN2+ diagnosed in either cervical biopsies or cone biopsy | at baseline ( within 3 months after index sample)
  The detection of underlying CIN2 or worse
The number of women with CIN2+ diagnosed in either cervical biopsies or cone biopsy | at follow-up ( 1.5 years after index sample)
  The detection of underlying CIN2 or worse
The number of women with CIN3+ diagnosed in either cervical biopsies or cone biopsy | at baseline ( within 3 months after index sample)
  The detection of underlying CIN3 or worse
The number of women with CIN3+ diagnosed in either cervical biopsies or cone biopsy | at follow-up (1.5 years after index sample)
  The detection of underlying CIN3 or worse

SECONDARY OUTCOMES:
Clinical accuracy (sensitivity and specificity of each triage marker and in different combinations) | at baseline (within 3 months after index sample)
  sensitivity to detect underlying CIN2+ and specificity to exclude underlying CIN2+
Clinical accuracy (sensitivity and specificity of each triage marker and in different combinations) | at follow-up (1.5 years after index sample)
  sensitivity to detect underlying CIN2+ and specificity to exclude underlying CIN2+
HPV genotype distribution | at baseline (within 3 months after index sample)
  We will measure the distribution of hrHPV types among these older women
DS positivity rate | at baseline (within 3 months after index sample)
  We will measure the DS positivity rate among these older women

CONTACTS AND LOCATIONS:
Overall Officials: mette tranberg, post doc, Principal Investigator — Randers Regional Hospital, Denmark
Locations (1):
- Department of Pathology, Randers, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
This is yet to be decided.